CLINICAL TRIAL: NCT03329976
Title: Validation of a Prognostic Score for Good Visual Recovery at One Year Following Combined Surgery for Cataract and Idiopathic Epiretinal Membrane
Acronym: PROCATMER
Status: Terminated | Type: Observational
Why Stopped: due to lack of recruitment
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: KAUFFMANN PHRCI 2016
Record Dates: First submitted 2017-10-13; First posted 2017-11-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Surgery for Cataract; Surgery for and Idiopathic Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: any person about to undergo combined surgery for cataract and ERM
  Interventions: Other: measurement of visual acuity

INTERVENTIONS:
Other: measurement of visual acuity — complete ophthalmologic examination of a macular SD-OCT, a fundus of eye, evaluation of the vision of contrasts (Pelli-Robson test) and quantification of metamorphopsies (M-Charts);

SUMMARY:
The prevalence of idiopathic epiretinal membranes (ERM) in people over 50 is estimated at 6 to 19%. Even though most cases show very few symptomats, they may induce alterations of the underlying retina and lead to visual impairment likely to greatly diminish quality of life in patients. Thanks to the ever-improving quality of vitreo-retinal surgery, ablation of these membranes is a frequent and safe procedure allowing a functional gain in the majority of cases. Given the increasing prevalence in the population concerned and the accelerated ageing of the lens after vitrectomy, cataract surgery is often associated with removal of the membrane. On the basis of a study in 142 patients, it was possible to identify clinical and morphological prognostic factors and to inclure them in a score to assess the chances of complete functional recovery at one year following the procedure . Age of the patient, the duration of symptoms, initial visual acuity and the quality of the junction between external and internal segments of photoreceptors in optic coherence tomography (OCT) appeared as significantly related to visual results. Using this score in a new prospective cohort would allow the investigators to make it a reliable and easy-to-use tool at the service of ophthalmologist surgeons and their patients and would provide scientific confirmation of the interest of earlier surgery in this disease. It would also allow the investigators to define in a validated and reproducible manner, a threshold for an ndication for ERM surgery, which is currently based on relatively subjective criteria mostly related to visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting idiopathic ERM visible on SD-OCT;
* Indication for combined cataract and ERM surgery in a context of a fall in visual acuity or disabling metamorphopsia;
* Patients who have provided verbal consent;
* Age ≥ 40 years.

Exclusion Criteria:

* Patients with secondary ERM (Diabetes WITH a history of diabetic retinopathy or maculopathy, occlusion of the retinal veins, uveitis intermediate/posterior uveitis or retinal tear/detachment in the studied eye;
* Patient présentant toute autre maculopathie ou neuropathie optique ;
* Patient presenting severe myopia (spherical equivalent ≥ 6 diopters or axial length ≥ 26 mm) ;
* Patients presenting any other ophthalmological disease independent of the ERM and likely to limit visual acuity
* Patients who have already undergone vitrectomy in the studied eye;
* Non-visible or poorly visible fundus due to a cloudy vitreous (Signal on OCT Cirrus <5, Quality score on OCT Spectralis < 20, signal trend index on OCT Optovue < 30)
* Patients without national health insurance cover
* Pregnant or breast-feeding women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any person about to undergo combined surgery for cataract and ERM
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
scale of monoyer at 5 meter | over the 12 months of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France